CLINICAL TRIAL: NCT05294939
Title: Randomized Clinical Trial to Analyze the Efficacy of Acute Intake of a Ketone Supplement on Performance in Professional Cross-country Road Cyclists
Brief Title: Efficacy of Acute Intake of Ketones on Performance in Professional Road Cyclists
Acronym: KETA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Católica San Antonio de Murcia (Other)
Responsible Party: Principal Investigator, Francisco Javier López Román, Principal Investigator, Universidad Católica San Antonio de Murcia
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: UCAMCFE-00022
Record Dates: First submitted 2022-01-10; First posted 2022-03-24 (Actual); Last update posted 2022-04-13 (Actual); Status verified 2021-11

CONDITIONS: Ketoses, Metabolic; Ketosis
MeSH Terms: conditions — Ketosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ketone monoester (Experimental): Consumption of 800mg/kg body weight of ketone monoester, divided in two intakes. The mixture will be prepared with bicarbonate. In addition, every hour they should consume 90g of carbohydrates.
  Interventions: Dietary Supplement: Ketone monoester
- Control product (Placebo Comparator): Consumption of placebo product (carbohydrates) masked with citric, divided in two intakes. The mixture will be prepared with bicarbonate. In addition, every hour they should consume 90g of carbohydrates.
  Interventions: Dietary Supplement: Control product consumption

INTERVENTIONS:
Dietary Supplement: Ketone monoester — Consumption of 800mg/kg body weight of ketone monoester, divided in two intakes. The mixture will be prepared with bicarbonate. In addition, every hour they should consume 90g of carbohydrates.
  Arms: Ketone monoester
Dietary Supplement: Control product consumption — Consumption of placebo product (carbohydrates) masked with citric, divided in two intakes. The mixture will be prepared with bicarbonate. In addition, 90g of carbohydrates should be consumed every hour.
  Arms: Control product

SUMMARY:
Randomized, controlled, double-blind, crossover clinical trial, depending on the product consumed, to analyze the efficacy on physical performance of a sports supplement consumed prior to and during competition or training.

DETAILED DESCRIPTION:
Subjects who meet the selection criteria will be randomly assigned to each of the study groups (investigational product or placebo, depending on the group to which they have been assigned). On the second day, participants will consume the product that subjects did not consume on the first day.

The product to be consumed will be ketone monoester. Participants will consume 800 mg/kg body weight, distributed in two intakes. The first one, half an hour before exercise and the same dose will be consumed one hour and a half after the first dose. The intakes will be accompanied by carbohydrates and bicarbonate.

The tests that the cyclists will perform are a time trial on a cycloergometer to measure performance, as well as a 30" sprint. Afterwards, the cyclists will do a 4 and a half hour training session at competition pace. After this training session, the participants will do the same time trial and the 30'' sprint.

ELIGIBILITY:
Inclusion Criteria:

* Male professional cyclists.
* Start the study with previous rest.

Exclusion Criteria:

* Participant suffering from chronic illness.
* Suffering a long-term injury that prevents her from training in the month prior to the intervention.
* Inability to understand the informed consent.
* Having consumed ketone bodies chronically in the previous four weeks.
* To have undergone cholecystectomy.

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2022-01-31 (Actual); Primary Completion 2022-02-05 (Actual); Study Completion 2022-03-28 (Actual)

PRIMARY OUTCOMES:
Physical performance | Change in performance after product consumption and training at a competitive level
  Measured using a power roller. Variables such as maximum power and average power

SECONDARY OUTCOMES:
Heart Rate | It will be measured on four different occasions. Two on the first day (after one intake of product and after a second intake and training at competitive pace) and 4 days later, the same measurements but with the opposite product.
  Measured by a chest strap
Microcapillary blood | It will be measured on four different occasions. Two on the first day (after one intake of product and after a second intake and training at competitive pace) and 4 days later, the same measurements but with the opposite product.
  This test provides biochemical variables (ABL90FLEX) with 70 ml of capillary blood.
Lactate | It will be measured on four different occasions. Two on the first day (after one intake of product and after a second intake and training at competitive pace) and 4 days later, the same measurements but with the opposite product.
  Lactate levels will be measured using the Lactate Pro
Ketone | It will be measured on four different occasions. Two on the first day (after one intake of product and after a second intake and training at competitive pace) and 4 days later, the same measurements but with the opposite product.
  Will be measured by the FreeStyle Optium
Blood glucose | It will be measured on four different occasions. Two on the first day (after one intake of product and after a second intake and training at competitive pace) and 4 days later, the same measurements but with the opposite product.
  Will be measured by the FreeStyle Optium
Blood glucose | It will be measured on a daily basis. Measurements will begin two days before the first performance test and end one day after the completion of the performance tests.
  It will be measured continuously by Supersapiens.
Heart rate variability | It will be measured every morning. Measurements will be started two days before the first performance test and finished one day after the end of the performance tests.
  It will be measured for 5 minutes upon awakening.
Stomach test | It will be measured on four different occasions. Two on the first day (after one intake of product and after a second intake and training at competitive pace) and 4 days later, the same measurements but with the opposite product.
  It will be measured by means of a visual analog scale from 0 to 10 to determine the annoyance produced by the product (0: none and 10: maximum annoyance).
Fatigue | It will be measured on four different occasions. Two on the first day (after one intake of product and after a second intake and training at competitive pace) and 4 days later, the same measurements but with the opposite product.
  Rate of perceived exertion

CONTACTS AND LOCATIONS:
Locations (1):
- Catholic University of Murcia, Murcia, Spain

IPD SHARING:
Plan to Share IPD: No